CLINICAL TRIAL: NCT05982275
Title: Anti-BCMA Chimeric Antigen Receptor (CARTemis-1) T-lymphocyte Therapy in the Treatment of Patients With Multiple Myeloma in Relapse After Allogeneic Transplant: Endothelial Growth Factor Receptor Expression as a Control Mechanism of Treatment-derived Complications
Brief Title: Trial of an Investigational Drug After Rejecting the Relapse of an Allogeneic Transplant
Acronym: CARTemis-1
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CARTemis-1
Record Dates: First submitted 2023-05-02; First posted 2023-08-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma; Allogeneic Stem Cell Transplantation
Keywords: Chimeric antigen receptor-T cell therapy; B-Cell Maturation Antigen
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARTemis-1 (Experimental): Dose escalation sequential cohorts CARTemis-1 will be self-administered intravenously one or two days, depending on the dose administered.
  Interventions: Genetic: CARTemis-1

INTERVENTIONS:
Genetic: CARTemis-1 — A dose escalation design will be applied in successive patient cohorts until identification of Dose Limiting Toxicity (maximum dose: 6x10^6 CAR-T/kg divided over 2 days).

SUMMARY:
Most patients with multiple myeloma (MM) die due to relapse resistant to current treatment, including treatment with anti-B cell maturation antigen (BCMA) CAR-T cells. To overcome some of the potential limitations of this therapy, a new and optimized Anti-BCMA CAR-T has been developed, with the aim of using it in patients with MM who relapse after Allogeneic Haematopoietic Haematopoietic Progenitor. This trial is a prospective phase I/II trial with a 3+3 design. Once Dose Limiting Toxicity is identified, Phase II will begin to assess the efficacy of the procedure.

DETAILED DESCRIPTION:
This trial is a prospective phase I/II trial with a 3+3 design. Once Dose Limiting Toxicity is identified (up to a maximum dose of 6x106 CAR-T/kg divided over 2 days), phase II of the trial will begin to assess the efficacy of the procedure.

A number of 25 patients will be included to evaluate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old with a diagnosis of post-allogeneic transplant relapse multiple myeloma.
2. Measurable disease at the time of screening
3. Previous treatment with ≥2 lines before and/or after allogeneic transplant.
4. Patients who are not receiving immunosuppressants at least 1 month before inclusion and who do not have active graft-versus-host disease.
5. Eastern Cooperative Oncology Group functional status from 0 to 1.
6. Life expectancy greater than 3 months (at the time of screening)
7. Patients who give their consent by signing the Informed Consent document.

Exclusion Criteria:

1. Active systemic immunosuppressive treatment
2. Patients who have previously received treatment with CAR-T Anti-BCMA.
3. Absolute lymphocyte count <0.2x109/L
4. Previous neoplasm, except if it has been in complete remission >3 years, with the exception of skin carcinoma (non-melanoma)
5. Active infection requiring treatment.
6. Active HIV, hepatitis B virus or hepatitis C virus infection.
7. Uncontrolled medical illness.
8. Severe organic disease that meets any of the following criteria: left ventricular ejection fraction <40%, carbon monoxide diffusion test <40%, glomerular filtration rate <50 ml/min, bilirubin >3 normal value (except Gilbert syndrome).
9. Previous diagnosis of symptomatic amyloid light chain or primary amyloidosis or POEMS Syndrome.
10. Pregnant or lactating women.
11. Women of childbearing age, unable or unwilling to use highly effective contraceptive methods.
12. Men who cannot or do not wish to use highly effective contraceptive methods. The partner of the male participants, if they are women of childbearing age, must also use highly effective contraceptive methods during the study period.
13. Contraindication to receive lymphodepleting chemotherapy.
14. Patients with known hypersensitivity to the active ingredients or any of the excipients of the product to be infused.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Purity of CARTemis-1 | Immediately after infusion
  Number of cases in which, after performing apheresis, the manufacturing process is completed and CARTemis-1 cells are infused
Maximum tolerated dose | Up to 30 days
  To determine the maximum tolerated dose of CarTemis-1
Infusion reactions | Immediately after intravenous administration of CARTemis-1
  To appearance of any of the following symptoms after intravenous administration of CARTemis-1: cardiac events, chills, dyspnea, fatigue, sudden hypertension, hypotension, nausea, pain, fever, skin rash, and urticaria.
Tumor lysis syndrome | Up to 30 days after treatment administration
  To increase nucleic acids, potassium, and phosphate in the blood
Serious Adverse Event | Up to 36 months after treatment administration
  Type, incidence, severity (graded by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0), timing, intensity, and relatedness of adverse events).
Suspected Unexpected Serious Adverse Reaction | Up to 36 months after treatment administration
  Describe the adverse event that occurs in a clinical trial subject, which is assessed by the sponsor and or study investigator as being unexpected, serious and as having a reasonable possibility of a causal relationship with the study drug.

SECONDARY OUTCOMES:
Number of Participants with cytopenias | During the first 90 days after administration of CARTemis-1
  Neutropenias or thrombopenias
Number of Participants with prolonged cytopenias | Up to 12 months after treatment administration
  Neutropenias or thrombopenias (grade ≥3) for more than 6 weeks
Duration of clinical response | Screening, day -5, -4, -3, +28, +56, +100 and months +4, +5, 6, +7, +8, +9, +10, +11, +12, +15 , +18, +21, +27, +30, +33, +36 or progression
  Duration of clinical response as assessed by Urinalysis (immunofixation, proteinuria and 24-h urine proteinogram), Blood tests (total immunoglobulin A, G and M, immunofixation and proteinogram (M component) in serum; serum free light chains), Bone Marrow Aspirate and Positron Emission Tomography.
Overall response rate | 3, 6 and 12 months after CARTemis-1 infusion
  Overall response rate as assessed by criteria of the International Myeloma Working Group
Time to complete remission | Up to 36 months after treatment administration
  Duration of clinical response as assessed by Urinalysis (immunofixation, proteinuria and 24-h urine proteinogram), Blood tests (total immunoglobulin A, G and M, immunofixation and proteinogram (M component) in serum; serum free light chains), Bone Marrow Aspirate and Positron Emission Tomography
Time to best response | Up to 36 months after treatment administration
  Duration of clinical response as assessed by Urinalysis (immunofixation, proteinuria and 24-h urine proteinogram), Blood tests (total immunoglobulin A, G and M, immunofixation and proteinogram (M component) in serum; serum free light chains), Bone Marrow Aspirate and Positron Emission Tomography
Negative Minimum Residual Disease Rate | 3, 6 and 12 months after CARTemis-1 infusion
  Residual amount of malignant cells in the bone marrow
Response rate of extramedullary disease | 3 months after CARTemis-1 infusion
  To measure of the metabolic activity of the human body by Positron Emission Tomography
Progression-free survival. | Up to 36 months after treatment administration
  Quantification of time between administration of CARTemis-1 and disease progression or death
Overall survival | Up to 36 months after treatment administration
  the time elapsed between the infusion of CARTemis-1 and the patient's death from any cause.
Persistence of CARTemis-1 | Peripheral blood:days 3,7,10,14,17 (only in cohort 3 and 4),21,30,56,90,128 and 156, and months 6,9,12,15,18,24 and relapse or month 36 post-infusion; Marrow: 1,3,6,12,18 and 24 months post-infusion and in the progression or month
  Presence of CARTemis-1 in peripheral blood and bone marrow
CART cell quality | During the manufacturing process, at the time of infusion and at Month+1, Month+3, Month+6, Month+12, Month+18 and Month+24 post-infusion
  Evaluation of the biological characteristics of CARTemis-1 performed by flow cytometry to identify the optimal time of expansion as well as to study the dynamics of CAR T cells during the manufacturing process and how the manufacturing impacts on CAR T cell features and, therefore, CAR T cell quality.
Expression of B cell maturation antigen (BCMA) | Screening and at the time of follow up when a relapse occurs, an average after 1 year
  Genetic expression of BCMA at selection and at relapse in patients
B cell maturation antigen (BCMA) levels | Screening, Day -5, Day 0, +1, +3, +7 y +28 and months +3, +6, +12, +18 and +24
  Serum soluble BCMA levels pre-treatment and during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Antonio Perez-Simon, MD-PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (5):
- Spain (5):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Complejo asistencial universitario de Salamanca, Salamanca
  - José Antonio Pérez Simón, Seville
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The results will be shared with the investigators involved in the study, and will be shared when the analysis of the results is performed.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Along the study
Access Criteria: Direct collaborators within the study